CLINICAL TRIAL: NCT02409329
Title: Improving Medication Adherence Among Underserved Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lindsay Mayberry, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 140562; 1R01DK100694-01A1 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-04-06 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REACH (Experimental): Participants will receive REACH text messages (individual-focused text messaging tailored to user's individual barriers to adherence and targeted to address other self-care behaviors) for 12 months.
  All participants will also receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: REACH; Behavioral: Helpline and A1c results
- REACH + FAMS (Experimental): In addition to the REACH text messages tailored to user's individual barriers to adherence, participants will receive FAMS components (monthly phone coaching and text messages supporting a goal set in coaching, plus the option to invite a family member/support person to receive text messages) for six months. After six months, participants in this arm will receive REACH text messages only.
  All participants will also receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: Helpline and A1c results; Behavioral: REACH + FAMS
- Helpline and A1c results (Active Comparator): Participants assigned to the control group will complete measures at each time point and maintain care as usual (i.e., medical treatment and physician monitoring).
  All participants will receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: Helpline and A1c results

INTERVENTIONS:
Behavioral: REACH — The intervention consists of daily text messaging tailored to user's individual barriers to medication adherence, text messages assessing user's adherence with feedback on progress, plus text messaging targeting other self-care behaviors.
  Arms: REACH
Behavioral: Helpline and A1c results — Participants complete study assessments, receive text messages advising how to access study A1c results, receive quarterly newsletters on healthy living with diabetes, and have access to a helpline for study- or diabetes medication-related questions.
Behavioral: REACH + FAMS — The intervention consists of REACH individually-focused text messaging, plus family-focused phone coaching session, goal-focused text messaging, and the option to invite a family member/support person to receive text messaging.
  Other Names: NCT02481596
  Arms: REACH + FAMS

SUMMARY:
This study evaluates a mobile phone-delivered intervention, called REACH (Rapid Education/Encouragement And Communications for Health), in supporting adults with type 2 diabetes in their self-management relative to a control group. The goal of this study is to determine if individually tailored content (based on the Information-Motivation-Behavioral Skills Model) delivered to the participant via text messages can improve the participant's glycemic control and adherence to diabetes medications. We will test whether our intervention improves adherence-related information, motivation, and behavioral skills and whether improving these mechanisms drives improvements in adherence and, in turn, glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Individuals who have received a diagnosis for type 2 diabetes mellitus
* Enrolled as a patient at a participating community health center
* Individuals currently being treated with oral and/or injectable diabetes medications

Exclusion Criteria:

* Non-English speakers
* Individuals who report they do not have a cell phone
* Individuals unwilling and/or not able to provide written informed consent
* Individuals with unintelligible speech (e.g., dysarthria)
* Individuals with a severe hearing or visual impairment
* Individuals who report a caregiver administers their diabetes medications Individuals who fail the cognitive screener administered during the baseline survey
* Individuals who cannot receive, read, and respond to a text after instruction from a trained research assistant
* Individuals whose most recent (within 12 months) HbA1c value was 6.8% or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay S Mayberry, MS, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Federally Qualified Health Centers and Vanderbilt Primary Care Clinics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be de-identified and made available following publication of the 15-month trial results to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after final trial results publication. No end date.
Access Criteria: Approval of a proposal by the study PI.

REFERENCES:
- [Background] Nelson LA, Mayberry LS, Wallston K, Kripalani S, Bergner EM, Osborn CY. Development and Usability of REACH: A Tailored Theory-Based Text Messaging Intervention for Disadvantaged Adults With Type 2 Diabetes. JMIR Hum Factors. 2016 Sep 8;3(2):e23. doi: 10.2196/humanfactors.6029. PMID 27609738
- [Background] Nelson LA, Wallston KA, Kripalani S, Greevy RA Jr, Elasy TA, Bergner EM, Gentry CK, Mayberry LS. Mobile Phone Support for Diabetes Self-Care Among Diverse Adults: Protocol for a Three-Arm Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 10;7(4):e92. doi: 10.2196/resprot.9443. PMID 29636319
- [Derived] Roddy MK, Mayberry LS, Nair D, Cavanaugh KL. Exploring mHealth potential to improve kidney function: secondary analysis of a randomized trial of diabetes self-care in diverse adults. BMC Nephrol. 2022 Aug 10;23(1):280. doi: 10.1186/s12882-022-02885-6. PMID 35948873
- [Derived] Mayberry LS, Bergner EM, Harper KJ, Laing S, Berg CA. Text messaging to engage friends/family in diabetes self-management support: acceptability and potential to address disparities. J Am Med Inform Assoc. 2019 Oct 1;26(10):1099-1108. doi: 10.1093/jamia/ocz091. PMID 31403688

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants were administratively withdrawn prior to randomization; 5 were unreachable during a pre-determined run-in period after enrollment, 1 behaved inappropriately with a research assistant during enrollment
Groups:
- REACH: Participants will receive REACH text messages (individual-focused text messaging tailored to user's individual barriers to adherence and targeted to address other self-care behaviors) for 12 months.
  All participants will also receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  REACH: The intervention consists of daily text messaging tailored to user's individual barriers to medication adherence, text messages assessing user's adherence with feedback on progress, plus text messaging targeting other self-care behaviors.
  Helpline and A1c results: Participants complete study assessments, receive text messages advising how to access study A1c results, receive quarterly newsletters on healthy living with diabetes, and have access to a helpline for study- or diabetes medication-related questions.
- REACH + FAMS: In addition to the REACH text messages tailored to user's individual barriers to adherence, participants will receive FAMS components (monthly phone coaching and text messages supporting a goal set in coaching, plus the option to invite a family member/support person to receive text messages) for six months. After 6 months, participants in this arm will receive REACH text messages only.
  All participants will also receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Helpline and A1c results: Participants complete study assessments, receive text messages advising how to access study A1c results, receive quarterly newsletters on healthy living with diabetes, and have access to a helpline for study- or diabetes medication-related questions.
  REACH + FAMS: The intervention consists of REACH individually-focused text mes
- Helpline and A1c Results: Participants assigned to the control group will complete measures at each time point and maintain care as usual (i.e., medical treatment and physician monitoring).
  All participants will receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Helpline and A1c results: Participants complete study assessments, receive text messages advising how to access study A1c results, receive quarterly newsletters on healthy living with diabetes, and have access to a helpline for study- or diabetes medication-related questions.
Period: Overall Study
Arm/Group | REACH | REACH + FAMS | Helpline and A1c Results
Started | 127 | 126 | 253
Completed | 122 | 120 | 244
Not Completed | 5 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- REACH + FAMS: In addition to the REACH text messages tailored to user's individual barriers to adherence, participants will receive FAMS components (monthly phone coaching and text messages supporting a goal set in coaching, plus the option to invite a family member/support person to receive text messages) for 6 months. After six months, participants in this arm will receive REACH text messages only.
  All participants will also receive text messages advising how to access their study A1c test results, receive quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Helpline and A1c results: Participants complete study assessments, receive text messages advising how to access study A1c results, receive quarterly newsletters on healthy living with diabetes, and have access to a helpline for study- or diabetes medication-related questions.
  REACH + FAMS: The intervention consists of REACH individually-focused text mes
- Total: Total of all reporting groups
Arm/Group | REACH | REACH + FAMS | Helpline and A1c Results | Total
Number analyzed (Participants) | 127 | 126 | 253 | 506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 97 | 206 | 412
  >=65 years | 18 | 29 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.4) | 55.7 (10.2) | 56.1 (9.4) | 55.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 135 | 274
  Male | 57 | 57 | 118 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 15 | 31
  Not Hispanic or Latino | 116 | 111 | 224 | 451
  Unknown or Not Reported | 3 | 7 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 4
  Asian | 3 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 51 | 49 | 98 | 198
  White | 64 | 63 | 128 | 255
  More than one race | 2 | 5 | 6 | 13
  Unknown or Not Reported | 6 | 6 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 127 | 126 | 253 | 506
Hemoglobin A1c (%) [Mean (Standard Deviation); unit: percent] | 8.72 (1.79) | 8.56 (1.90) | 8.53 (1.80) | 8.58 (1.82)
Medication Adherence - Summary of Diabetes Self-Care Activities medication subscale [Mean (Standard Deviation); unit: days in a week] — as measured by the Summary of Diabetes Self-Care Activities (SDSCA) Medications subscale; response options are days in the last week ranging from 0 to 7, with 7 representing perfect adherence
  days in a week | 6.25 (1.37) | 6.37 (1.09) | 6.41 (1.16) | 6.36 (1.20)
Medication Adherence - Adherence to Refills and Medications Scale for Diabetes [Mean (Standard Deviation); unit: score on a scale] — as measured by the Adherence to Refills and Medications Scale for Diabetes (ARMS-D); reverse coded such that higher scores indicate better adherence on a scale from 11 to 44
  score on a scale | 39.90 (3.74) | 39.66 (3.54) | 40.21 (3.34) | 39.99 (3.54)
Use of dietary information - Personal Diabetes Questionnaire [Mean (Standard Deviation); unit: score on a scale] — as measured by the Personal Diabetes Questionnaire diet subscale "Use of information for decision making"; possible range 1-6, higher indicates more use of dietary information (better)
  score on a scale | 3.09 (1.74) | 2.85 (1.57) | 2.96 (1.70) | 2.97 (1.68)
Problem eating behaviors - Personal Diabetes Questionnaire [Mean (Standard Deviation); unit: score on a scale] — Personal Diabetes Questionnaire diet subscale "Problem eating behavior"; possible range 1-6 with higher indicating more problem eating behavior (worse)
  score on a scale | 3.23 (1.08) | 3.43 (1.04) | 3.35 (1.16) | 3.34 (1.11)
MET-minutes per week - International Physical Activity Questionnaire-short form [Mean (Standard Deviation); unit: MET-minutes per week] — as measured by International Physical Activity Questionnaire-Short form [metabolic equivalent minutes (MET-minutes) per week] where more MET-minutes per week indicates more physical activity
  MET-minutes per week | 2565.11 (3108.48) | 1836.23 (2183.39) | 2348.91 (2853.58) | 2274.58 (2777.96)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycemic Control as Indicated by Hemoglobin A1c (HbA1c)
Description: as measured by Hemoglobin A1c (%) with higher values indicating worse glycemic control and an improvement of 0.5% considered clinically meaningful
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: We compared participants receiving the REACH intervention (combining REACH and REACH + FAMS) with participants not receiving REACH (in condition Helpline and A1c Results).
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
percent
  3 months | 8.29 (1.49) | 8.59 (1.65)
  6 months | 8.32 (1.65) | 8.57 (2.15)
  12 months | 8.66 (1.97) | 8.70 (2.10)
  15 months | 8.59 (1.81) | 8.61 (1.95)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; Any REACH vs. Helpline and A1c results. We used generalized estimating equations (GEE) with a working-exchangeable correlation structure and identity link, adjusting for baseline and allowing a time-treatment interaction. For the HbA1c model, we allowed for a three-way interaction between time, treatment group, and baseline HbA1c because there was descriptive evidence that the effect was modified by baseline HbA1c values. Multiply imputed data (m=1,000) using chained equations; Test type: Superiority — We performed an omnibus test of the treatment effect at 3 and 6 months using a robust variance-covariance based Wald statistic. We used ordinary least squares linear regression with Huber-White heteroscedasticity-consistent standard errors to obtain point estimates and 95% CIs for the intervention effect at each time; p = .0493, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = -0.313, 95% CI 2-sided [-0.610 to -0.017] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — We performed an omnibus test of the treatment effect at 3, 6, 12, and 15 months using a robust variance-covariance based Wald statistic. We used ordinary least squares linear regression with Huber-White heteroscedasticity-consistent standard errors to obtain point estimates and 95% CIs for the intervention effect at each time; p = 0.260, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = -0.070, 95% CI 2-sided [-0.380 to 0.240] — 15-month point estimate

2. Secondary Outcome: Change in Self-reported Medication Adherence
Description: as measured by the Summary of Diabetes Self-Care Activities (SDSCA) Medications subscale; response options are days in the last week ranging from 0 to 7, with 7 representing perfect adherence
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
days per week
  3 months | 6.59 (0.96) | 6.38 (1.25)
  6 months | 6.64 (0.89) | 6.24 (1.51)
  12 months | 6.50 (1.09) | 6.27 (1.46)
  15 months | 6.36 (1.22) | 6.18 (1.45)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; Any REACH vs. Helpline and A1c results. We used generalized estimating equations with a working-exchangeable correlation structure and identity link, adjusting for baseline and allowing a time-treatment interaction. Multiply imputed data (m=1,000) using chained equations; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .001, Wald statistic — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.406, 95% CI 2-sided [0.196 to 0.615] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.003, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.210, 95% CI 2-sided [-0.031 to 0.450] — 15-month point estimate

3. Secondary Outcome: Change in Self-reported Medication Adherence
Description: as measured by the Adherence to Refills and Medications Scale for Diabetes (ARMS-D); reverse coded such that higher scores indicate better adherence on a scale from 11 to 44
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
score on a scale
  3 months | 40.4 (3.62) | 40.4 (3.45)
  6 months | 40.6 (3.48) | 40.2 (3.49)
  12 months | 40.3 (3.48) | 40.2 (3.99)
  15 months | 40.5 (3.24) | 40.4 (3.90)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; Any REACH vs. Helpline and A1c results. We used generalized estimating equations (GEE) with a working-exchangeable correlation structure and identity link, adjusting for baseline and allowing a time-treatment interaction. Multiply imputed data (m=1,000) using chained equations; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.376, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.540, 95% CI 2-sided [-0.012 to 1.090] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.434, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.278, 95% CI 2-sided [-0.319 to 0.875] — 15-month point estimate

4. Other Pre Specified Outcome: Change in Adherence to Dietary Behavior
Description: as measured by the Personal Diabetes Questionnaire diet subscale "Use of information for decision making"; possible range 1-6, higher indicates more use of dietary information (better)
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
score on a scale
  3 months | 3.17 (1.59) | 2.84 (1.58)
  6 months | 3.34 (1.56) | 2.93 (1.62)
  12 months | 3.22 (1.58) | 2.88 (1.61)
  15 months | 3.17 (1.65) | 3.01 (1.77)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0012, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.399, 95% CI 2-sided [0.160 to 0.637] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.003, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.152, 95% CI 2-sided [-0.121 to 0.426] — 15-month point estimate

5. Other Pre Specified Outcome: Change in Adherence to Dietary Behavior
Description: Personal Diabetes Questionnaire diet subscale "Problem eating behavior"; possible range 1-6 with higher indicating more problem eating behavior (worse)
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
score on a scale
  3 months | 3.17 (1.03) | 3.28 (1.13)
  6 months | 3.11 (0.95) | 3.18 (1.06)
  12 months | 3.09 (1.07) | 3.13 (1.09)
  15 months | 3.18 (1.15) | 3.18 (1.11)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.632, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = -0.061, 95% CI 2-sided [-0.218 to 0.095] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.572, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 0.005, 95% CI 2-sided [-0.202 to 1.100] — 15-month point estimate

6. Other Pre Specified Outcome: Change in Physical Activity
Description: as measured by International Physical Activity Questionnaire-Short form [metabolic equivalent minutes (MET-minutes) per week] where more MET-minutes per week indicates more physical activity
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MET-minutes per week
Arm/Group | REACH | Helpline and A1c Results
Number analyzed (Participants) | 253 | 253
MET-minutes per week
  3 months | 2285 (2973) | 2139 (2501)
  6 months | 2332 (3168) | 1991 (2547)
  12 months | 2573 (3329) | 2273 (2883)
  15 months | 2221 (2973) | 2239 (2774)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.703, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 369, 95% CI 2-sided [-142 to 881] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.465, GEE, Wald test — A priori threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); Predicted mean difference = 26, 95% CI 2-sided [-459 to 511] — 15-month point estimate

7. Other Pre Specified Outcome: Change in Glycemic Control - REACH Only vs. Control & REACH+FAMS vs. Control
Description: as measured by hemoglobin A1c (HbA1c, %) We may be under-powered to for these comparative analyses.
Time Frame: Baseline, 3 months, 6 months, 12 months, 15 months
Population: We compared participants receiving the REACH intervention only with those receiving REACH + FAMS and with participants not receiving REACH (in condition Helpline and A1c Results). This analysis was subsetted to participants with baseline HbA1c greater than or equal to 8.5% with the goal of improved power.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | REACH | REACH + FAMS | Helpline and A1c Results
Number analyzed (Participants) | 59 | 52 | 106
percent
  3 months | 9.12 (1.41) | 8.98 (1.61) | 9.47 (1.77)
  6 months | 8.88 (1.64) | 9.14 (1.53) | 9.74 (2.37)
  12 months | 9.45 (1.89) | 9.57 (2.19) | 9.67 (2.21)
  15 months | 9.28 (1.97) | 9.41 (1.74) | 9.57 (2.25)
Statistical Analysis 1: Comparison: REACH vs Helpline and A1c Results; To evaluate if REACH only and REACH+FAMS had similar effects on HbA1c relative to control, we subsetted to participants with baseline HbA1c greater than or equal to 8.5% to maximize our power for these analyses. We used generalized estimating equations (GEE) with a working-exchangeable correlation structure and identity link, adjusting for baseline and allowing a time-treatment interaction. Multiply imputed data (m=1,000) using chained equations; Test type: Superiority — Testing superiority of REACH only relative to control. We used ordinary least squares linear regression with Huber-White heteroscedasticity-consistent standard errors to obtain point estimates and 95% CIs for the intervention effect at each time; Predicted mean difference = -0.75, 95% CI 2-sided [-1.38 to -0.12] — 6-month point estimate
Statistical Analysis 2: Comparison: REACH vs Helpline and A1c Results; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — [test comment as in outcome 7, analysis 1]; Predicted mean difference = -0.31, 95% CI 2-sided [-1.00 to 0.39] — 12-month point estimate
Statistical Analysis 3: Comparison: REACH + FAMS vs Helpline and A1c Results; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Testing superiority of REACH_FAMS relative to control. We used ordinary least squares linear regression with Huber-White heteroscedasticity-consistent standard errors to obtain point estimates and 95% CIs for the intervention effect at each time; Predicted mean difference = -0.65, 95% CI 2-sided [-1.26 to -0.05] — 6-month point estimate
Statistical Analysis 4: Comparison: REACH + FAMS vs Helpline and A1c Results; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Testing superiority of REACH+FAMS relative to control. We used ordinary least squares linear regression with Huber-White heteroscedasticity-consistent standard errors to obtain point estimates and 95% CIs for the intervention effect at each time; Predicted mean difference = -0.31, 95% CI 2-sided [-0.96 to 0.51] — 12-month point estimate

ADVERSE EVENTS:
Time Frame: We followed participants for 15 months of study participation, lasting from recruitment start May 2016 until the last participant completed 15-month follow-up in June 2019.
Arm/Group | REACH | REACH + FAMS | Helpline and A1c Results
All-Cause Mortality (participants affected / at risk) | 3/127 | 2/126 | 3/253
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/126 | 0/253
Other Adverse Events (participants affected / at risk) | 0/127 | 0/126 | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT02409329/SAP_000.pdf
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT02409329/Prot_001.pdf